CLINICAL TRIAL: NCT06765161
Title: Efgartigimod in IVIG Dependent Myasthenia Gravis Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Clinique Neuro-Outaouais (Other)
Collaborators: argenx (Industry)
Responsible Party: Principal Investigator, Dr. Francois Jacques, Neurologist, Clinique Neuro-Outaouais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-CA-NEU-96
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Myasthaenia Gravis
Keywords: Myasthenia gravis; Vyvgart; IVIG
MeSH Terms: conditions — Myasthenia Gravis | interventions — efgartigimod alfa

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment (Experimental): Efgartigimod infusion
  Interventions: Drug: efgartigimod administration

INTERVENTIONS:
Drug: efgartigimod administration — efgartigimod infusion
  Other Names: Vyvgart

SUMMARY:
This study is an open label, single center, prospective, 26 weeks study with descriptive analysis where IVIG is replaced by efgartigimod therapy. MG-ADL and MGQOL evaluations will occur weekly throughout the study to week 26.

DETAILED DESCRIPTION:
Objectives:

To determine if efgartigimod is equivalent or non-inferior in efficacy to IVIG in the treatment of stable, acetylcholine receptor antibody positive, IVIG dependent myasthenia gravis patients.

To determine patient treatment preference between IVIG and efgartigimod in stable, IVIG dependent acetylcholine receptor antibody positive myasthenia gravis patients.

To determine the safety and tolerability of efgartigimod administered in a fixed regular dosing regimen over 6 months in stable IVIG dependent acetylcholine receptor antibody positive myasthenia gravis patients.

IVIG will be discontinued one week prior to the baseline visit (week 0) while other concurrent medications (non-steroidal immunosuppressive therapies (NSISTs), acetylcholinesterase (AChE) inhibitors or corticosteroids) for myasthenia will be kept unchanged for the duration of the study. The dose and frequency of efgartigimod treatment will be 10mg/kg (max of 1200mg) administered as a one-hour intravenous infusion every week x 4 infusions followed by a four-week break and repeated for a total four treatment cycles till week 24 and then followed by a two-week observation with an end of study visit at week 26.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed informed consent. 2. Age 18-80 years 3. Acetylcholine receptor antibody positive, myasthenia gravis patients, with stable disease for the past four or more months. Stable disease is defined as no change in dosage or interval in IVIG treatments and without any significant change in clinical status.

  4. No modification or addition of NSISTs in the past six months 5. No modification or addition in corticosteroid therapy for the past three months 6. Myasthenia Gravis diagnosis was supported by abnormal neurotransmission test or history of improvement with AChE inhibitors.

  7. Receiving chronic regular IVIG treatments for myasthenia gravis for the past year or more.

Exclusion Criteria:

* 1. Patients with previous rituxan or eculizumab treatment or plasma exchange within the past six months 2. Patients with previous thymectomy within the past 3months 3. Patients that have active Hepatitis B, are seropositive for Hepatitis C or HIV or have latent, untreated or active TB or any other significant active infection 4. Patients that have at screening a serum IgG less than 6.0gm/L or a history of chronic hypogammaglobulinemia from any cause.

  5. Patients that are pregnant or considering becoming pregnant in the next 6 months.

  6. Patients with severe renal impairment (eGFR less than 30ml/min) 7. Patients who in the opinion of the investigator should not participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2027-01-06 (Estimated)

PRIMARY OUTCOMES:
MG-ADL | a sustained decrease persistent for at least 4 consecutive weeks over the 26 week period
  The percentage of patients who do not experience, at any time during the study, a 2 or more-point deterioration from their averaged baseline MG-ADL score that is sustained for a period of 4 or more consecutive weeks. (stable or improved patients)

SECONDARY OUTCOMES:
QMG | those who experience a sustained decrease for 4 consecutive weeks during the 26 week period
  The percentage of patients who do not experience, at any time during the study, a 3 or more-point deterioration from their baseline QMG score that is sustained for a period of 4 or more consecutive weeks. (stable or improved patients)
MGQOL | during the whole study period of 26 weeks
  The change in group, mean MGQOL score from the averaged baseline to the week 26 end of study visit.
incidence of patients who are still receiving efgartigimod by the end of the 26 weeks | for the duration of the 26 week study
  incidence of patients who are still receiving efgartigimod by the end of the 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: François Jacques, Doctor, Principal Investigator — Clinique Neuro-Outaouais
Locations (1):
- Clinique Neuro-Outaouais, Gatineau, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burns TM, Sadjadi R, Utsugisawa K, Gwathmey KG, Joshi A, Jones S, Bril V, Barnett C, Guptill JT, Sanders DB, Hobson-Webb L, Juel VC, Massey J, Gable KL, Silvestri NJ, Wolfe G, Cutter G, Nagane Y, Murai H, Masuda M, Farrugia ME, Carmichael C, Birnbaum S, Hogrel JY, Nafissi S, Fatehi F, Ou C, Liu W, Conaway M. International clinimetric evaluation of the MG-QOL15, resulting in slight revision and subsequent validation of the MG-QOL15r. Muscle Nerve. 2016 Dec;54(6):1015-1022. doi: 10.1002/mus.25198. Epub 2016 Nov 7. PMID 27220659
- [Background] Barnett C, Katzberg H, Nabavi M, Bril V. The quantitative myasthenia gravis score: comparison with clinical, electrophysiological, and laboratory markers. J Clin Neuromuscul Dis. 2012 Jun;13(4):201-5. doi: 10.1097/CND.0b013e31824619d5. PMID 22622164
- [Background] Howard JF Jr, Bril V, Vu T, Karam C, Peric S, De Bleecker JL, Murai H, Meisel A, Beydoun SR, Pasnoor M, Guglietta A, Van Hoorick B, Steeland S, T'joen C, Utsugisawa K, Verschuuren J, Mantegazza R; ADAPT+ Study Group. Long-term safety, tolerability, and efficacy of efgartigimod (ADAPT+): interim results from a phase 3 open-label extension study in participants with generalized myasthenia gravis. Front Neurol. 2024 Jan 17;14:1284444. doi: 10.3389/fneur.2023.1284444. eCollection 2023. PMID 38318236
- [Background] Wolfe GI, Herbelin L, Nations SP, Foster B, Bryan WW, Barohn RJ. Myasthenia gravis activities of daily living profile. Neurology. 1999 Apr 22;52(7):1487-9. doi: 10.1212/wnl.52.7.1487. PMID 10227640
- [Background] Howard JF Jr, Bril V, Vu T, Karam C, Peric S, Margania T, Murai H, Bilinska M, Shakarishvili R, Smilowski M, Guglietta A, Ulrichts P, Vangeneugden T, Utsugisawa K, Verschuuren J, Mantegazza R; ADAPT Investigator Study Group. Safety, efficacy, and tolerability of efgartigimod in patients with generalised myasthenia gravis (ADAPT): a multicentre, randomised, placebo-controlled, phase 3 trial. Lancet Neurol. 2021 Jul;20(7):526-536. doi: 10.1016/S1474-4422(21)00159-9. PMID 34146511
- [Background] Sesarman A, Vidarsson G, Sitaru C. The neonatal Fc receptor as therapeutic target in IgG-mediated autoimmune diseases. Cell Mol Life Sci. 2010 Aug;67(15):2533-50. doi: 10.1007/s00018-010-0318-6. Epub 2010 Mar 9. PMID 20217455